CLINICAL TRIAL: NCT04209465
Title: MasterKey-01: A Phase 1/2, Open-label, Two-part, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics & Antitumor Activity of BDTX-189, an Inhibitor of Allosteric ErbB Mutations, in Patients w/ Advanced Solid Malignancies
Brief Title: A Study of BDTX-189, an Orally Available Allosteric ErbB Inhibitor, in Patients With Advanced Solid Tumors.
Acronym: MasterKey-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The development of BDTX-189 was discontinued by the sponsor.
Sponsor: Black Diamond Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BDTX-189-01
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor
Keywords: solid tumor; HER2 mutation; exon 20 insertion mutation; HER2 positive; Genes, HER2; Genes, erbb2; HER2 amplification; HER2 overexpression; genes, exon 20 insertion; lung cancer; non-small cell lung cancer; breast cancer; colon cancer; colorectal cancer; bladder cancer; endometrial cancer; gastric cancer; biliary tract cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Colonic Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms; Endometrial Neoplasms; Stomach Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 - Dose escalation (Experimental): In Part A, cohorts of patients with select HER2, HER3, or EGFR alterations received increasing doses of BDTX-189.
  Interventions: Drug: BDTX-189

INTERVENTIONS:
Drug: BDTX-189 — Participants received a daily, oral dose of BDTX-189 as part of a 3 week cycle.

SUMMARY:
This was a clinical study with an orally administered drug, BDTX-189 in participants with advanced solid tumors that had select mutations or alterations in human epidermal growth factor receptor 2 (HER2/ErbB2) genes or epidermal growth factor receptor (EGFR/ErbB1). The main goals of this study were to:

* Find the recommended dose of BDTX-189 that can be given safely to participants
* Learn more about the side effects of BDTX-189
* Learn what the body does to BDTX-189 after it has been taken (pharmacokinetics or PK)
* Determine the preliminary antitumor activity of BDTX-189 in participants with select allosteric ErbB gene mutations

DETAILED DESCRIPTION:
BDTX-189 is an irreversible, small molecular inhibitor that is highly selective versus wild-type EGFR and potent for cancer driver mutations of the ErbB family, including extracellular, transmembrane, and kinase domain allosteric mutations of HER2, as well as EGFR and HER2 exon 20 insertion mutations. These allosteric ErbB mutations are found in 1 - 2 % of most solid tumors and enriched in some cancers with a prevalence of about 2 - 7% such as in non-small cell lung cancer, breast cancer, colorectal cancer, bladder cancer, and endometrial cancer. Currently approved HER2 and EGFR directed therapies are not active against the spectrum of allosteric mutations at relevant and tolerated exposure levels.

This Phase 1/2 multi-center, open-label trial was a first-in-human study that evaluated BDTX-189 orally administered daily as a single agent in patients with solid tumors harboring select mutations or alterations. The Phase 1 portion was a dose escalation primarily designed to assess the safety and tolerability of BDTX-189 and to determine a recommended Phase 2 dose (RP2D). Phase 1 focused on patients with a solid tumor and with alterations such as:

* Allosteric HER2 or HER3 mutation(s)
* EGFR or HER2 exon 20 insertion mutation(s)
* HER2 amplified or overexpressing tumors
* EGFR exon 19 deletion or L858R mutation

Eligible mutations must have been determined by a validated next-generation sequencing (NGS) test routinely used by each institution and performed in a CLIA-certified or equivalent laboratory.

The Phase 2 portion was not initiated.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically- or cytologically-confirmed locally advanced or metastatic solid tumor with documented recurrence or disease progression from standard anticancer therapy in the advanced/metastatic setting
* No standard therapy available or standard therapy is considered unsuitable or intolerable according to the Investigator and consultation with the Medical Monitor

Phase 1 Only:

* Solid tumor patients with alterations that may be associated with antitumor activity based on preclinical data for BDTX-189 such as:

  1. Allosteric HER2 or HER3 mutation(s)
  2. EGFR or HER2 exon 20 insertion mutation(s)
  3. HER2 amplified or overexpressing tumors
  4. EGFR exon 19 deletion or L858R mutation

Eligible mutations must be determined by a validated next-generation sequencing (NGS) test routinely used by each institution and performed in a CLIA-certified or equivalent laboratory.

* Adequate archival tumor tissue or willing to undergo pretreatment biopsy
* Measurable disease according to RECIST version 1.1

Main Exclusion Criteria:

* Clinical laboratory values meeting the following criteria within 4 weeks (28 days) prior to baseline:

  1. Serum creatinine ≥1.5 × upper limit of normal (ULN) or calculated creatinine clearance ≤60 mL/min using Cockcroft-Gault equation
  2. Total bilirubin ≥1.5 × ULN or ≥3.0 × ULN in the presence of documented Gilbert's syndrome
  3. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2.5 × ULN, or AST or ALT ≥5.0 × ULN in the presence of liver metastases
  4. Hematologic function:

     1. Absolute neutrophil count (ANC) ≤1000 cells/μL
     2. Hemoglobin ≤8.5 g/dL or 5.28 mmol/L
     3. Platelet count ≤75,000/μL
* Significant cardiovascular disease, including:

  1. Cardiac failure New York Heart Association Class III or IV, or left ventricular ejection fraction (LVEF) <50% or below the lower limit of the Institution's normal range
  2. Myocardial infarction, severe or unstable angina within 6 months prior to baseline
  3. Significant thrombotic or embolic events within 3 months prior to baseline
  4. History or presence of any uncontrolled cardiovascular disease
  5. Personal or family history of long QT syndrome
* ECG findings meeting any of the following criteria:

  1. Evidence of second- or third-degree atrioventricular block
  2. Clinically significant arrhythmia (as determined by the Investigator)
  3. QTcF interval of >470 msec
* Leptomeningeal or untreated and/or symptomatic CNS malignancies (primary or metastatic)
* Women who are pregnant or breast-feeding
* Taking or unable to discontinue proton pump inhibitors within 1 week prior to baseline
* Known concurrent KRAS mutation
* Known tumor-harboring resistance mutations including EGFR T790M or C797S mutations or HER2 C805S mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (24):
  - 9250, Scottsdale, Arizona
  - 9405, Long Beach, California
  - 9474, Orange, California
  - 7141, New Haven, Connecticut
  - 4080, Lake Mary, Florida
  - 4100, Orlando, Florida
  - 9535, Plantation, Florida
  - 4060, Sarasota, Florida
  - 9035, Atlanta, Georgia
  - 9530, Rolling Meadows, Illinois
  - 9092, New Orleans, Louisiana
  - 9203, Boston, Massachusetts
  - 9209, Buffalo, New York
  - 9215, New York, New York
  - 9236, New York, New York
  - 9264, Portland, Oregon
  - 7122, Pittsburgh, Pennsylvania
  - 4107, Chattanooga, Tennessee
  - 3000, Nashville, Tennessee
  - 9003, Dallas, Texas
  - 9117, Houston, Texas
  - 9538, Webster, Texas
  - 9112, Fairfax, Virginia
  - 9173, Milwaukee, Wisconsin
- 9500, Copenhagen, Denmark
- France (5):
  - 9501, Bordeau
  - 9525, Lille
  - 9373, Lyon
  - 9512, Poitiers
  - 9476, Rennes
- Spain (8):
  - 9496, Barcelona
  - 9363, Barcelona
  - 9508, Barcelona
  - 9429, Madrid
  - 9495, Madrid
  - 9383, Madrid
  - 9382, Madrid
  - 9510, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erika Paige Hamilton, Manish R. Patel, Jordi Rodon, David S. Hong, Alison M. Schram, Pasi A. Janne, Patricia LoRusso, Jasgit C. Sachdev, Sai Hong Ou, Elizabeth A Buck, Matthew O'Connor, Nigel Waters, Karsten Witt, Carl Cook. Masterkey-01: Phase I/II, open-label multicenter study to assess safety, tolerability, pharmacokinetics, and antitumor activity of BDTX-189, an inhibitor of allosteric ErbB mutations, in patients with advanced solid malignancies. J Clin Oncol 38: 2020 (suppl; abstr TPS3665)

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation 25 mg QD: Patients who received doses at 25 mg once daily under fasted conditions.
- Dose Escalation 50 mg QD: Patients who received doses at 50 mg once daily under fasted conditions.
- Dose Escalation 100 mg QD: Patients who received doses at 100 mg once daily under fasted conditions.
- Dose Escalation 200 mg QD: Patients who received doses at 200 mg once daily under fasted conditions.
- Dose Escalation 400 mg QD: Patients who received 400 mg once daily under fasted conditions.
- Dose Escalation 800 mg QD: Patients who received 800 mg once daily under fasted conditions.
- Dose Escalation 800 mg QD Not Fasted: Patients who received 800 mg once daily under not fasted conditions.
- Dose Escalation 1000 mg QD: Patients who received 1000 mg once daily under fasted condition.
- Dose Escalation 1200 mg QD: Patients who received 1200 mg once daily under fasted conditions.
- Dose Escalation 400 mg BID: Patients who received 400 mg twice daily under not fasted conditions.
- Dose Escalation 600 mg BID: Patients who received 600 mg twice daily under not fasted conditions.
- Dose Escalation 800 mg BID: Patients who received 800 mg twice daily under fasted conditions.
- Phase 1 Safety Expansion: Patients who received 800 mg once daily as a safety expansion group under not fasted conditions.
Period: Overall Study
Arm/Group | Dose Escalation 25 mg QD | Dose Escalation 50 mg QD | Dose Escalation 100 mg QD | Dose Escalation 200 mg QD | Dose Escalation 400 mg QD | Dose Escalation 800 mg QD | Dose Escalation 800 mg QD Not Fasted | Dose Escalation 1000 mg QD | Dose Escalation 1200 mg QD | Dose Escalation 400 mg BID | Dose Escalation 600 mg BID | Dose Escalation 800 mg BID | Phase 1 Safety Expansion
Started | 1 | 1 | 1 | 2 | 10 | 18 | 13 | 7 | 6 | 4 | 6 | 5 | 17
Completed | 0 (Study was discontinued prematurely) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 1
Not Completed | 1 | 1 | 1 | 2 | 10 | 16 | 10 | 6 | 6 | 4 | 5 | 5 | 16
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 2 | 7 | 2 | 2 | 1 | 1 | 1 | 0 | 10
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 1 | 2 | 8 | 5 | 3 | 4 | 1 | 3 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Started new therapy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated early by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation 800 mg QD NF: Patients who received 800 mg once daily under not fasted conditions.
- Dose Escalation 1000 mg QD: Patients who received 1000 mg once daily under not fasted conditions
- Safety Expansion 800 mg QD: Patients in safety expansion who received 800 mg once daily under not fasted conditions.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation 25 mg QD | Dose Escalation 50 mg QD | Dose Escalation 100 mg QD | Dose Escalation 200 mg QD | Dose Escalation 400 mg QD | Dose Escalation 800 mg QD | Dose Escalation 800 mg QD NF | Dose Escalation 1000 mg QD | Dose Escalation 1200 mg QD | Dose Escalation 400 mg BID | Dose Escalation 600 mg BID | Dose Escalation 800 mg BID | Safety Expansion 800 mg QD | Total
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 10 | 18 | 13 | 7 | 6 | 4 | 6 | 5 | 17 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 1 | 4 | 9 | 10 | 4 | 6 | 0 | 4 | 5 | 7 | 52
  >=65 years | 0 | 1 | 0 | 1 | 6 | 9 | 3 | 3 | 0 | 4 | 2 | 0 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 | 65 | 51 | 60 (17.0) | 64.5 (9.48) | 65.4 (11.94) | 60.2 (7.00) | 61.4 (7.00) | 55.8 (6.59) | 71.0 (6.06) | 59.3 (11.99) | 58.0 (5.70) | 65.3 (10.34) | 63.1 (10.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 5 | 9 | 9 | 4 | 6 | 3 | 5 | 3 | 8 | 54
  Male | 1 | 0 | 1 | 1 | 5 | 9 | 4 | 3 | 0 | 1 | 1 | 2 | 9 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 5 | 12
  Not Hispanic or Latino | 1 | 1 | 1 | 2 | 9 | 15 | 11 | 6 | 4 | 4 | 4 | 5 | 11 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 2 | 10 | 18 | 13 | 7 | 6 | 4 | 6 | 5 | 12 | 86
  Spain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities as a Determinant of the Recommended Phase 2 Dose (RP2D)
Description: Certain toxicities will be considered dose-limiting unless clearly attributable to an extraneous cause, such as underlying disease.
Time Frame: After the first dose of treatment for up to 21 days.
Population: DLT-Evaluable
Measure: Number; unit: participants
Groups:
- 25 mg QD: Patients who received doses at 25 mg once daily under fasted conditions.
- 50 mg QD: Patients who received doses at 50 mg once daily under fasted conditions.
- 100 mg QD: Patients who received doses at 100 mg once daily under fasted conditions.
- 200 mg QD: Patients who received doses at 200 mg once daily under fasted conditions.
- 400 mg QD: Patients dosed at 400 mg once daily under fasted conditions
- 800 mg QD Fasted: Patients enrolled at 800 mg once daily under fasted conditions
- 800 mg QD Not Fasted: Patients enrolled at 800 mg once daily under not fasted conditions
- 1000 mg QD: Patients enrolled at 1000 mg once daily under not fasted conditions
- 1200 mg QD: Patients enrolled at 1200 mg once daily under fasted conditions
- 400 mg BID: Patients enrolled at 400 mg twice daily under not fasted conditions
- 600 mg BID: Patients enrolled at 600 mg twice daily under not fasted conditions
- 800 mg BID: Patients enrolled at 800 mg twice daily under fasted conditions
- Safety Expansion Set 800 mg QD: Safety expansion group patients enrolled at 800 mg once daily under not fasted conditions.
Arm/Group | 25 mg QD | 50 mg QD | 100 mg QD | 200 mg QD | 400 mg QD | 800 mg QD Fasted | 800 mg QD Not Fasted | 1000 mg QD | 1200 mg QD | 400 mg BID | 600 mg BID | 800 mg BID | Safety Expansion Set 800 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 10 | 18 | 13 | 7 | 6 | 4 | 6 | 5 | 17
participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 3 | 3 | 1

2. Secondary Outcome: Phase 1: Incidence of Treatment-emergent Adverse Events as a Measure of Safety and Tolerability of BDTX-189
Description: Adverse events will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Time Frame: From Cycle 1 Day 1 (each cycle is 21 days) until 30 days post last dose
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg QD | 50 mg QD | 100 mg QD | 200 mg QD | 400 mg QD | 800 mg QD Fasted | 800 mg QD Not Fasted | 1000 mg QD | 1200 mg QD | 400 mg BID | 600 mg BID | 800 mg BID | Safety Expansion Set 800 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 10 | 18 | 13 | 7 | 6 | 4 | 6 | 5 | 17
Participants | 0 | 0 | 0 | 2 | 10 | 18 | 13 | 7 | 6 | 4 | 6 | 5 | 17

3. Secondary Outcome: Phase 1: Plasma Concentration of BDTX-189 as a Measure of Pharmacokinetics
Description: Blood samples will be taken to measure the plasma concentrations of BDTX-189 in both a fed and fasted state.
Time Frame: Multiple time points during Cycles 1-4 (each cycle is 21 days)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per mililiter (ng/mL)
Arm/Group | Dose Escalation 25 mg QD | Dose Escalation 50 mg QD | Dose Escalation 100 mg QD | Dose Escalation 200 mg QD | Dose Escalation 400 mg QD | Dose Escalation 800 mg QD | Dose Escalation 800 mg QD NF | Dose Escalation 1000 mg QD | Dose Escalation 1200 mg QD | Dose Escalation 400 mg BID | Dose Escalation 600 mg BID | Dose Escalation 800 mg BID | Safety Expansion 800 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 9 | 13 | 11 | 1 | 3 | 3 | 2 | 3 | 22
Nanogram per mililiter (ng/mL) | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) is not calculable for a single participant. | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) is not calculable for a single participant. | NA (NA) — Geometric Mean (Geometric Coefficient of Variation) is not calculable for a single participant. | 151 (67.5) | 170 (104) | 268 (72.7) | 341 (46.4) | 0 (0) | 352 (77.8) | 123 (133) | 84.5 (39) | 165 (53.8) | 248 (77.8)

4. Secondary Outcome: Phase 1: Objective Response Rate as a Preliminary Measure of Antitumor Activity
Description: Objective response is defined as the proportion of participants who achieved a complete response (CR; disappearance of all target and non-target lesions) or partial response (PR; at least a 30% decrease from baseline in the sum of diameters of target lesions) per RECIST version 1.1.
Time Frame: Assessed until disease progression or death for up to 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation 1000 mg QD: Patients who received 1000 mg once daily under fasted conditions.
- Safety Expansion 800 mg QD: Safety expansion patients who received 800 mg once daily under not fasted conditions.
Arm/Group | Dose Escalation 25 mg QD | Dose Escalation 50 mg QD | Dose Escalation 100 mg QD | Dose Escalation 200 mg QD | Dose Escalation 400 mg QD | Dose Escalation 800 mg QD | Dose Escalation 800 mg QD NF | Dose Escalation 1000 mg QD | Dose Escalation 1200 mg QD | Dose Escalation 400 mg BID | Dose Escalation 600 mg BID | Dose Escalation 800 mg BID | Safety Expansion 800 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 10 | 18 | 13 | 7 | 6 | 4 | 6 | 5 | 17
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Stable disease (SD) | 0 | 1 | 1 | 0 | 4 | 9 | 3 | 0 | 1 | 2 | 4 | 1 | 7
  Non-complete response/non-partial response (non-CR/non-PR) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Progressive disease (PD) | 1 | 0 | 0 | 2 | 6 | 4 | 5 | 3 | 2 | 1 | 2 | 3 | 8
  Not evaluable (NE) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 2 | 1 | 0 | 1 | 2

5. Secondary Outcome: Phase 1: Progression-free Survival as a Measure of Antitumor Activity
Description: Progression-free survival is the time from first study dose until disease progression (PD; target lesion increase of 20% and at least 5mm from smallest on-study lesion sum, the appearance of new lesions, or unequivocal progression of non-target lesions) per RECIST v1.1.
Time Frame: Assessed until disease progression or death for up to 12 months
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Dose Escalation 25 mg QD | Dose Escalation 50 mg QD | Dose Escalation 100 mg QD | Dose Escalation 200 mg QD | Dose Escalation 400 mg QD | Dose Escalation 800 mg QD | Dose Escalation 800 mg QD NF | Dose Escalation 1000 mg QD | Dose Escalation 1200 mg QD | Dose Escalation 400 mg BID | Dose Escalation 600 mg BID | Dose Escalation 800 mg BID | Safety Expansion 800 mg QD
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 10 | 18 | 13 | 7 | 6 | 4 | 6 | 5 | 17
Months | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 1.61 [0.941 to 2.279] | 1.866 [0.909 to 2.115] | 2.306 [0.493 to 4.143] | 5.158 [0.502 to 11.122] | 1.416 [1.147 to 2.189] | 1.572 [0.429 to 2.819] | 1.508 [0.688 to 2.327] | 2.252 [1.434 to 3.482] | 1.354 [0.548 to 2.160] | 1.772 [1.428 to 3.592]

ADVERSE EVENTS:
Time Frame: Patients remained on-study (on-treatment) until progression, adverse event, or withdrawal of consent. Mean duration of treatment across all dose levels was 11.7 months (median was 6.6 months).
Groups:
- Dose Escalation 800 mg QD NF: Patients who received 800 mg once daily under not fasted (NF) conditions.
- Safety Expansion 800 mg QD: Safety expansion group of patients who received 800 mg once daily under not fasted conditions.
Arm/Group | Dose Escalation 25 mg QD | Dose Escalation 50 mg QD | Dose Escalation 100 mg QD | Dose Escalation 200 mg QD | Dose Escalation 400 mg QD | Dose Escalation 800 mg QD | Dose Escalation 800 mg QD NF | Dose Escalation 1000 mg QD | Dose Escalation 1200 mg QD | Dose Escalation 400 mg BID | Dose Escalation 600 mg BID | Dose Escalation 800 mg BID | Safety Expansion 800 mg QD
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 0/2 | 2/10 | 7/18 | 2/13 | 2/7 | 1/6 | 1/4 | 1/6 | 0/5 | 10/17
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 2/2 | 2/10 | 8/18 | 1/13 | 1/7 | 1/6 | 1/4 | 2/6 | 3/5 | 4/17
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 2/2 | 10/10 | 18/18 | 13/13 | 7/7 | 6/6 | 4/4 | 6/6 | 5/5 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation 25 mg QD (N=1) | Dose Escalation 50 mg QD (N=1) | Dose Escalation 100 mg QD (N=1) | Dose Escalation 200 mg QD (N=2) | Dose Escalation 400 mg QD (N=10) | Dose Escalation 800 mg QD (N=18) | Dose Escalation 800 mg QD NF (N=13) | Dose Escalation 1000 mg QD (N=7) | Dose Escalation 1200 mg QD (N=6) | Dose Escalation 400 mg BID (N=4) | Dose Escalation 600 mg BID (N=6) | Dose Escalation 800 mg BID (N=5) | Safety Expansion 800 mg QD (N=17)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasogenic cerebral edema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation 25 mg QD (N=1) | Dose Escalation 50 mg QD (N=1) | Dose Escalation 100 mg QD (N=1) | Dose Escalation 200 mg QD (N=2) | Dose Escalation 400 mg QD (N=10) | Dose Escalation 800 mg QD (N=18) | Dose Escalation 800 mg QD NF (N=13) | Dose Escalation 1000 mg QD (N=7) | Dose Escalation 1200 mg QD (N=6) | Dose Escalation 400 mg BID (N=4) | Dose Escalation 600 mg BID (N=6) | Dose Escalation 800 mg BID (N=5) | Safety Expansion 800 mg QD (N=17)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 12 (12) | 9 (9) | 5 (5) | 4 (4) | 4 (4) | 5 (5) | 5 (5) | 12 (12)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 10 (10) | 8 (8) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 3 (3) | 10 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 9 (9) | 4 (4) | 4 (4) | 5 (5) | 2 (2) | 3 (3) | 3 (3) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 7 (7)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 7 (7) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Edema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Large intestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early. Phase 2 was not conducted. Limited data collection was performed for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT04209465/Prot_SAP_000.pdf